CLINICAL TRIAL: NCT03853122
Title: Effect of a Common Exercise Programme With an Individualized Progression Criterion Based on the Measurement of Neuromuscular Capacity Versus Eccentric Training for Lower Limb Tendinopathies (MaLaGa Trial): Randomised Clinical Trial
Brief Title: Exercise With Individual Dosage Against the Best Current Practice in Lower Limb Tendinopathy (MaLaGa Trial)
Acronym: MaLaGa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Director, Clinical Research, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DOSIS&TENDON
Record Dates: First submitted 2019-02-11; First posted 2019-02-25 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-05

CONDITIONS: Tendinopathy
Keywords: tendinopathy; exercise; dosage; physiotherapy
MeSH Terms: conditions — Tendinopathy; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, with two parallel groups (control and intervention)
Who Masked: Outcomes Assessor
Masking Description: Assessors are not aware of the allocation group of the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best current practice exercise programme (Active Comparator): Therapeutic physical exercise, best current practice:
  Achilles tendinopathy: ALFREDSON ECCENTRIC PROTOCOL: two exercises performed eccentrically, twice daily, 7 days/week, 14 weeks (6 weeks are added to the program to match the volume of weeks of the experimental group).
  Patellar tendinopathy: ALFREDSON ECCENTRIC PROTOCOL: one exercise performed eccentrically, twice daily, 7 days/week, 14 weeks (6 weeks are added to the program to match the volume of weeks of the experimental group).
  Gluteal Tendinopathy: EXERCISE LEAP PROTOCOL, from daily to twice weekly, 14 weeks (6 weeks are added to the program to match the volume of weeks of the experimental group).
  Interventions: Other: Best current practice exercise programme
- Experimental exercise programme (Experimental): Therapeutic physical exercise common for the three locations (Achilles, patellar and gluteal tendinopathy), based on an individual dosage and neuromuscular adaptations (five stages):
  Strength training four exercises, once daily, three times/week, 14 weeks Aerobic training: Once daily, twice weekly
  Interventions: Other: Experimental exercise programme

INTERVENTIONS:
Other: Best current practice exercise programme — Therapeutic Physical Exercise programme based on the protocol of Afredson (for Achilles and patellar tendinopathies) and LEAP (for gluteal tendinopathy).
  Achilles tendinopathy: ALFREDSON ECCENTRIC PROTOCOL: 3 sets of 15 repetitions of two eccentric exercises
  Patellar tendinopathy: ALFREDSON ECCENTRIC PROTOCOL: 3 sets of 15 repetions of one eccentric exercise
  Gluteal Tendinopathy: EXERCISE LEAP PROTOCOL: an exercise programme divided into stages with progression in different exercises, volumes and loads
  Other Names: Alfredson protocol; LEAP protocol
  Arms: Best current practice exercise programme
Other: Experimental exercise programme — Therapeutic Physical Exercise programme structured in five stages oriented to specific neuromuscular adaptations based on the characteristics of the neuromuscular system, once daily, three times/week, sets, repetitions and load based on individually performed tests.
  Other Names: MaLaGa protocol
  Arms: Experimental exercise programme

SUMMARY:
This study compares the effect of a therapeutic physical exercise programme based on an individualized control of the exercise dose by monitoring the force-speed curves against the current best practice in the treatment of tendinopathies of the lower limb. Half of the participants will receive the experimental intervention, while the other half will receive the best current practice.

DETAILED DESCRIPTION:
The current best practice is based on a progressive strength training sustained in the continuous model of tendinopathy proposed by Cook and Purdam (Cook & Purdam, 2009), showing in the literature this methodology more effective than the wait and see approach or that the use of corticosteroid injections, accentuating the differences in long-term follow-up evaluations (Mellor et al., 2018). However, the current system lacks an objectification methodology for the severity of the pathology and objective criteria for the progression of the load, usually based on subjective feelings of discomfort or pre-established intensities.

Therefore, the investigators hypothesize that the development and introduction of a methodology for the quantification and progression of the loads, with an individual control and management of the exercise dose, as well as the execution of specific exercises for each one of them, could improve the clinica and functional results. Moreover, achieving neuromuscular adaptations based on the characteristics of the neuromuscular system, could improve the times and results of the intervention, as well as the rate of treatment failures, in the tendinopathies of the lower limbs.

ELIGIBILITY:
Inclusion Criteria:

1. People between 18 and 65 years with a clinical diagnosis of mid-portion Achilles, patellar, or gluteal tendinopathy;
2. Pain duration for at least one month.

Exclusion Criteria:

1. Corticosteroid injection in the studied tendon in the last 12 months;
2. Other injuries in the affected lower limb in the last 12 months;
3. Previous surgery for musculoskeletal causes of the affected lower limb in the last 12 months;
4. Tendinous rupture history in the affected lower limb;
5. Systemic diseases such as rheumatic arthritis or diabetes mellitus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Victorian Institute of Sport Assessment (VISA) questionnaire POST | Post, 14 weeks after start of the intervention (when intervention is finished)
  Visa-A for Achilles tendon, Visa-P for Patellar tendon, Visa-G for Gluteal tendon: functional mobility, life participation, and pain. Assessed from 0 (worst value) to 100 (best value).

SECONDARY OUTCOMES:
Victorian Institute of Sport Assessment (VISA) questionnaire PRE | Baseline, 1 week before start of the intervention
  Visa-A model for Achilles tendon, Visa-P model for Patellar tendon, Visa-G model for Gluteal tendon: functional mobility, life participation, and pain. Assessed from 0 (worst value) to 100 (best value).
Victorian Institute of Sport Assessment (VISA) questionnaire SHOR TERM | Short term, 7 weeks after start of the intervention
  Visa-A for Achilles tendon, Visa-P for Patellar tendon, Visa-G for Gluteal tendon: functional mobility, life participation, and pain. Assessed from 0 (worst value) to 100 (best value).
Victorian Institute of Sport Assessment (VISA) questionnaire Follow-up | 52 weeks after the start of the intervention
  Visa-A for Achilles tendon, Visa-P for Patellar tendon, Visa-G for Gluteal tendon: functional mobility, life participation, and pain. Assessed from 0 (worst value) to 100 (best value).
Central Sensitization Inventory (CSI) PRE | Baseline, 1 week before start of the intervention
  Questionnaire to help identify patients with Central Sensitivity Syndromes. Range 0-100. Five severity levels developed to help aid in the clinical interpretation of the CSI (subclinical = 0-29; mild = 30-39; moderate = 40-49; severe = 50-59; and extreme = 60-100)
Central Sensitization Inventory (CSI) SHORT TERM | Short term, 7 weeks after start of the intervention
  Questionnaire to help identify patients with Central Sensitivity Syndromes. Range 0-100. Five severity levels developed to help aid in the clinical interpretation of the CSI (subclinical = 0-29; mild = 30-39; moderate = 40-49; severe = 50-59; and extreme = 60-100)
Central Sensitization Inventory (CSI) POST | Post, 14 weeks after start of the intervention (when intervention is finished)
  Questionnaire to help identify patients with Central Sensitivity Syndromes. Range 0-100. Five severity levels developed to help aid in the clinical interpretation of the CSI (subclinical = 0-29; mild = 30-39; moderate = 40-49; severe = 50-59; and extreme = 60-100)
Central Sensitization Inventory (CSI) FOLLOW-UP | 52 weeks after start of the intervention
  Questionnaire to help identify patients with Central Sensitivity Syndromes. Range 0-100. Five severity levels developed to help aid in the clinical interpretation of the CSI (subclinical = 0-29; mild = 30-39; moderate = 40-49; severe = 50-59; and extreme = 60-100)
Örebro Musculoskeletal Pain Questionnaire (ÖMPQ) PRE | Baseline, 1 week before start of the intervention
  OMPSQ is a self-administered pain screening questionnaire applied to identify patients with acute or subacute musculoskeletal pain who are at risk of delayed recovery. A higher score indicates a higher disability. The maximum score is 210 points; a score of < 105 points indicates a low disability, that between 105 and 130 points indicates a moderate disability and that > 130 points indicates a high disability
Örebro Musculoskeletal Pain Questionnaire (ÖMPQ) SHORT TERM | Short term, 7 weeks after start of the intervention
  OMPSQ is a self-administered pain screening questionnaire applied to identify patients with acute or subacute musculoskeletal pain who are at risk of delayed recovery. A higher score indicates a higher disability. The maximum score is 210 points; a score of < 105 points indicates a low disability, that between 105 and 130 points indicates a moderate disability and that > 130 points indicates a high disability
Örebro Musculoskeletal Pain Questionnaire (ÖMPQ) POST | Post, 14 weeks after start of the intervention (when intervention is finished)
  OMPSQ is a self-administered pain screening questionnaire applied to identify patients with acute or subacute musculoskeletal pain who are at risk of delayed recovery. A higher score indicates a higher disability. The maximum score is 210 points; a score of < 105 points indicates a low disability, that between 105 and 130 points indicates a moderate disability and that > 130 points indicates a high disability
Örebro Musculoskeletal Pain Questionnaire (ÖMPQ) FOLLOW-UP | 52 weeks after start of the intervention
  OMPSQ is a self-administered pain screening questionnaire applied to identify patients with acute or subacute musculoskeletal pain who are at risk of delayed recovery. A higher score indicates a higher disability. The maximum score is 210 points; a score of < 105 points indicates a low disability, that between 105 and 130 points indicates a moderate disability and that > 130 points indicates a high disability
Fear Avoidance Components Scale (FACS) PRE | Baseline, 1 week before start of the intervention
  The FACS scale comprehensively assesses the presence of fear avoidance beliefs and attitudes in people with painful medical conditions. The FACS instructions ask participants to reflect on past painful experiences, and to indicate the degree to which these experiences influence on their activity. There are 20 thoughts or feelings related to avoidance, on 6-point scales with the end points (0) completely disagree and (5) completely agree. The FACS yields a total score between 0, best score, and 100, worst score.
Fear Avoidance Components Scale (FACS) SHORT TERM | Short term, 7 weeks after start of the intervention
  The FACS scale comprehensively assesses the presence of fear avoidance beliefs and attitudes in people with painful medical conditions. The FACS instructions ask participants to reflect on past painful experiences, and to indicate the degree to which these experiences influence on their activity. There are 20 thoughts or feelings related to avoidance, on 6-point scales with the end points (0) completely disagree and (5) completely agree. The FACS yields a total score between 0, best score, and 100, worst score.
Fear Avoidance Components Scale (FACS) POST | Post, 14 weeks after start of the intervention (when intervention is finished)
  The FACS scale comprehensively assesses the presence of fear avoidance beliefs and attitudes in people with painful medical conditions. The FACS instructions ask participants to reflect on past painful experiences, and to indicate the degree to which these experiences influence on their activity. There are 20 thoughts or feelings related to avoidance, on 6-point scales with the end points (0) completely disagree and (5) completely agree. The FACS yields a total score between 0, best score, and 100, worst score.
Fear Avoidance Components Scale (FACS) FOLLOW-UP | 52 weeks after start of the intervention
  The FACS scale comprehensively assesses the presence of fear avoidance beliefs and attitudes in people with painful medical conditions. The FACS instructions ask participants to reflect on past painful experiences, and to indicate the degree to which these experiences influence on their activity. There are 20 thoughts or feelings related to avoidance, on 6-point scales with the end points (0) completely disagree and (5) completely agree. The FACS yields a total score between 0, best score, and 100, worst score.
European Quality of Life-5 Dimensions (EQ-5D) PRE | Baseline, 1 week before start of the intervention
  EQ-5D is a standardized instrument for measuring generic health status. The EQ-5D questionnaire has two components: health state description and evaluation. In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. Each dimension is rated in 5 levels from "I have no problem with..." to "I am unable to..."
European Quality of Life-5 Dimensions (EQ-5D) SHORT TERM | Short term, 7 weeks after start of the intervention
  EQ-5D is a standardized instrument for measuring generic health status. The EQ-5D questionnaire has two components: health state description and evaluation. In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. Each dimension is rated in 5 levels from "I have no problem with..." to "I am unable to..."
European Quality of Life-5 Dimensions (EQ-5D) POST | Post, 14 weeks after start of the intervention (when intervention is finished)
  EQ-5D is a standardized instrument for measuring generic health status. The EQ-5D questionnaire has two components: health state description and evaluation. In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. Each dimension is rated in 5 levels from "I have no problem with..." to "I am unable to..."
European Quality of Life-5 Dimensions (EQ-5D) FOLLOW-UP | 52 weeks after start of the intervention
  EQ-5D is a standardized instrument for measuring generic health status. The EQ-5D questionnaire has two components: health state description and evaluation. In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. Each dimension is rated in 5 levels from "I have no problem with..." to "I am unable to..."
Lower Limb Functional Index (LLFI) PRE | Baseline, 1 week before start of the intervention
  The LLFI is an index designed for assessing the functional capacity of the lower limbs with a combination of constructs that includes body functions, body structures, activities and participation, and environmental factors. The LLFI has 25 phrases as items and participants have to select which ones they identify with. The final score is calculated with the following formula: 100 - (number of sentences chosen x 4). The LLFI yields a total score (between 100, best score, and 0, worst score).
Lower Limb Functional Index (LLFI) POST | Post, 14 weeks after start of the intervention (when intervention is finished)
  The LLFI is an index designed for assessing the functional capacity of the lower limbs with a combination of constructs that includes body functions, body structures, activities and participation, and environmental factors. The LLFI has 25 phrases as items and participants have to select which ones they identify with. The final score is calculated with the following formula: 100 - (number of sentences chosen x 4). The LLFI yields a total score (between 100, best score, and 0, worst score).
Lower Limb Functional Index (LLFI) SHORT TERM | Short term, 7 weeks after start of the intervention
  The LLFI is an index designed for assessing the functional capacity of the lower limbs with a combination of constructs that includes body functions, body structures, activities and participation, and environmental factors. The LLFI has 25 phrases as items and participants have to select which ones they identify with. The final score is calculated with the following formula: 100 - (number of sentences chosen x 4). The LLFI yields a total score (between 100, best score, and 0, worst score).
Lower Limb Functional Index (LLFI) FOLLOW-UP | 52 weeks after start of the intervention
  The LLFI is an index designed for assessing the functional capacity of the lower limbs with a combination of constructs that includes body functions, body structures, activities and participation, and environmental factors. The LLFI has 25 phrases as items and participants have to select which ones they identify with. The final score is calculated with the following formula: 100 - (number of sentences chosen x 4). The LLFI yields a total score (between 100, best score, and 0, worst score).
Lower limb Strength PRE | Short term, 7 weeks after start of the intervention
  Assessment of the isometric strength in the leg press machine using a s-beam load cell
Lower limb Strength SHORT TERM | Short term, 7 weeks after start of the intervention
  Assessment of the isometric strength in the leg press machine using a s-beam load cell
Lower limb Strength POST | Post, 14 weeks after start of the intervention (when intervention is finished)
  Assessment of the isometric strength in the leg press machine using a s-beam load cell
Lower limb Strength FOLLOW-UP | 52 weeks after start of the intervention
  Assessment of the isometric strength in the leg press machine using a s-beam load cell
Muscular Thickness PRE | Baseline, 1 week before start of the intervention
  Measurement of the muscular thickness (in cm) by Ultrasonography
Muscular Thickness SHORT TERM | Short term, 7 weeks after start of the intervention
  Measurement of the muscular thickness (in cm) by Ultrasonography
Muscular Thickness POST | Post, 14 weeks after start of the intervention (when intervention is finished)
  Measurement of the muscular thickness (in cm) by Ultrasonography
Muscular Thickness FOLLOW-UP | 52 weeks after start of the intervention
  Measurement of the muscular thickness (in cm) by Ultrasonography
Pressure Pain Threshold PRE | Baseline, 1 week before start of the intervention
  Measurement of the Pressure Pain Threshold of tendon with a hand-held algometer. The tester is placed perpendicular to the skin over the test area, increasing the pressure 30kPa/s. Participants are instructed to indicate when the sensation change from comfortable pressure to slightly unpleasant pain. Test is repeated three times with one minute of rest between repetitions. The mean value is used for the analysis.
Pressure Pain Threshold SHORT TERM | Short term, 7 weeks after start of the intervention
  Measurement of the Pressure Pain Threshold of tendon with a hand-held algometer. The tester is placed perpendicular to the skin over the test area, increasing the pressure 30kPa/s. Participants are instructed to indicate when the sensation change from comfortable pressure to slightly unpleasant pain. Test is repeated three times with one minute of rest between repetitions. The mean value is used for the analysis.
Pressure Pain Threshold POST | Post, 14 weeks after start of the intervention (when intervention is finished)
  Measurement of the Pressure Pain Threshold of tendon with a hand-held algometer. The tester is placed perpendicular to the skin over the test area, increasing the pressure 30kPa/s. Participants are instructed to indicate when the sensation change from comfortable pressure to slightly unpleasant pain. Test is repeated three times with one minute of rest between repetitions. The mean value is used for the analysis.
Pressure Pain Threshold FOLLOW-UP | 52 weeks after start of the intervention
  Measurement of the Pressure Pain Threshold of tendon with a hand-held algometer. The tester is placed perpendicular to the skin over the test area, increasing the pressure 30kPa/s. Participants are instructed to indicate when the sensation change from comfortable pressure to slightly unpleasant pain. Test is repeated three times with one minute of rest between repetitions. The mean value is used for the analysis.
Pain at rest measured with Visual Analogue Scale (VAS) PRE | Baseline, 1 week before start of the intervention
  Measurement of the Pain at rest with a 100 mm VAS scale, 0 being no pain and 100 being the worst imaginable pain
Pain at rest measured with Visual Analogue Scale (VAS) SHORT TERM | Short term, 7 weeks after start of the intervention
  Measurement of the Pain at rest with a 100 mm VAS scale, 0 being no pain and 100 being the worst imaginable pain
Pain at rest measured with Visual Analogue Scale (VAS) POST | Post, 14 weeks after start of the intervention (when intervention is finished)
  Measurement of the Pain at rest with a 100 mm VAS scale, 0 being no pain and 100 being the worst imaginable pain
Pain at rest measured with Visual Analogue Scale (VAS) FOLLOW UP | 52 weeks after start of the intervention
  Measurement of the Pain at rest with a 100 mm VAS scale, 0 being no pain and 100 being the worst imaginable pain
Pain during activity (running) measured with Visual Analogue Scale (VAS) PRE | Baseline, 1 week before start of the intervention
  Measurement of the Pain during activity (running) with a 100 mm VAS scale, 0 being no pain and 100 being the worst imaginable pain
Pain during activity (running) measured with Visual Analogue Scale (VAS) SHORT-TERM | Short term, 7 weeks after start of the intervention
  Measurement of the Pain during activity (running) with a 100 mm VAS scale, 0 being no pain and 100 being the worst imaginable pain
Pain during activity (running) measured with Visual Analogue Scale (VAS) POST | Post, 14 weeks after start of the intervention (when intervention is finished)
  Measurement of the Pain during activity (running) with a 100 mm VAS scale, 0 being no pain and 100 being the worst imaginable pain
Pain during activity (running) measured with Visual Analogue Scale (VAS) FOLLOW UP | 52 weeks after start of the intervention
  Measurement of the Pain during activity (running) with a 100 mm VAS scale, 0 being no pain and 100 being the worst imaginable pain
Treatment satisfaction PRE | Baseline, 1 week before start of the intervention
  Treatment satisfaction assessed using a visual analog scale, from 0 to 100mm, with 0 being "not at all satisfied" and 10 being "extremely satisfied".
Treatment satisfaction SHORT-TERM | Short term, 7 weeks after start of the intervention
  Treatment satisfaction assessed using a visual analog scale, from 0 to 100mm, with 0 being "not at all satisfied" and 10 being "extremely satisfied".
Treatment satisfaction POST | Post, 14 weeks after start of the intervention (when intervention is finished)
  Treatment satisfaction assessed using a visual analog scale, from 0 to 100mm, with 0 being "not at all satisfied" and 10 being "extremely satisfied".
Treatment satisfaction FOLLOW UP | 52 weeks after start of the intervention
  Treatment satisfaction assessed using a visual analog scale, from 0 to 100mm, with 0 being "not at all satisfied" and 10 being "extremely satisfied".
Lower limb Strength measured with hand-held dinamometer PRE | Baseline, 1 week before start of the intervention
  Lower limb Strength measured with hand-held dinamometer (ankle plantarflexion for Achilles tendinopathy, knee extension for patellar tendinopathy, and hip abduction for gluteal tendinopathy). Two repetitions are performed and the mean value is used for the analysis.
Lower limb Strength measured with hand-held dinamometer POST | Post, 14 weeks after start of the intervention (when intervention is finished)
  Lower limb Strength measured with hand-held dinamometer (ankle plantarflexion for Achilles tendinopathy, knee extension for patellar tendinopathy, and hip abduction for gluteal tendinopathy). Two repetitions are performed and the mean value is used for the analysis.
Lower limb Strength measured with hand-held dinamometer SHORT TERM | Short term, 7 weeks after start of the intervention
  Lower limb Strength measured with hand-held dinamometer (ankle plantarflexion for Achilles tendinopathy, knee extension for patellar tendinopathy, and hip abduction for gluteal tendinopathy). Two repetitions are performed and the mean value is used for the analysis.
Lower limb Strength measured with hand-held dinamometer FOLLOW UP | 52 weeks after start of the intervention
  Lower limb Strength measured with hand-held dinamometer (ankle plantarflexion for Achilles tendinopathy, knee extension for patellar tendinopathy, and hip abduction for gluteal tendinopathy). Two repetitions are performed and the mean value is used for the analysis.
HDEMG profile with Non Invasive Surface High-Density Electromyography (HDEMG) PRE | Baseline, 1 week before start of the intervention
  Non invasive surface HDEMG during maximal isometric voluntary contraction performed in a leg press machine. Surface HDEMG is recorded during 20 seconds. Data obtained is analysed to extract the mean discharge rate of the motor units (in fires per second) and the recruitment and derecruitment threshold (in Nw). This variable will only be assessed in a randomly selected subgroup of each arm.
HDEMG profile with Non Invasive Surface High-Density Electromyography (HDEMG) POST | Post, 14 weeks after start of the intervention (when intervention is finished)
  Non invasive surface HDEMG during maximal isometric voluntary contraction performed in a leg press machine. Surface HDEMG is recorded during 20 seconds. Data obtained is analysed to extract the mean discharge rate of the motor units (in fires per second) and the recruitment and derecruitment threshold (in Nw). This variable will only be assessed in a randomly selected subgroup of each arm.
Amount of physical activity with International Physical Activity Questionnaire Short Form (IPAQ-SF) | Baseline, 1 week before start of the intervention
  Amount of physical activity of the patients through seven questions about the physical activity performed the previous seven days. Physical activity can be interpreted as a numerical value (reported as median MET-minutes) and as low, moderate, or high activity levels.
Amount of physical activity with International Physical Activity Questionnaire Short Form (IPAQ-SF) | Short term, 7 weeks after start of the intervention
  Amount of physical activity of the patients through seven questions about the physical activity performed the previous seven days. Physical activity can be interpreted as a numerical value (reported as median MET-minutes) and as low, moderate, or high activity levels.
Amount of physical activity with International Physical Activity Questionnaire Short Form (IPAQ-SF) | Post, 14 weeks after start of the intervention (when intervention is finished)
  Amount of physical activity of the patients through seven questions about the physical activity performed the previous seven days. Physical activity can be interpreted as a numerical value (reported as median MET-minutes) and as low, moderate, or high activity levels.
Amount of physical activity with International Physical Activity Questionnaire Short Form (IPAQ-SF) | 52 weeks after start of the intervention
  Amount of physical activity of the patients through seven questions about the physical activity performed the previous seven days. Physical activity can be interpreted as a numerical value (reported as median MET-minutes) and as low, moderate, or high activity levels.

REFERENCES:
- [Derived] Escriche-Escuder A, Cuesta-Vargas AI, Casana J. Effect of a common exercise programme with an individualised progression criterion based on the measurement of neuromuscular capacity versus current best practice for lower limb tendinopathies (MaLaGa trial): a protocol for a randomised clinical trial. BMJ Open. 2021 Aug 17;11(8):e046729. doi: 10.1136/bmjopen-2020-046729. PMID 34404699